CLINICAL TRIAL: NCT05574907
Title: Accuracy and Safety of 68Ga-FAPI PET/CT in the Diagnosis of Axillary Lymph Node Metastasis in Early Breast Cancer Patients: A Prospective Cohort Study
Brief Title: Characterizing Breast Cancer With 68Ga-FAPI PET/CT (PFB-01)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PekingUMCH-FAPI-BC-1
Record Dates: First submitted 2022-10-07; First posted 2022-10-12 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 68Ga-FAPI PET/CT (Experimental): Inject 68Ga-FAPI and then perform PET/CT scan.
  Interventions: Diagnostic Test: 68Ga-FAPI PET/CT scan

INTERVENTIONS:
Diagnostic Test: 68Ga-FAPI PET/CT scan — Patients with suspected breast cancer underwent 68Ga-FAPI PET/CT after an injection of 74-148 MBq (2-4 mCi) 68Ga-FAPI to image lesions of breast cancer.

SUMMARY:
Fibroblast activation protein (FAP) is overexpressed in cancer-associated fibroblasts (CAFs), which constitute a major proportion of cells within the tumor microenvironment, especially in breast cancer. 68Ga-FAPI has been developed as a tumor-targeting agent. This prospective study is going to investigate the performance and value of 68Ga-FAPI PET/CT in patients with breast cancer.

DETAILED DESCRIPTION:
Breast cancer is a complex, heterogeneous disease comprising numerous distinct biological subtypes characterized by variant pathobiological features and clinical behaviors. 18F-fluorodeoxyglucose (18F-FDG) PET/CT, an essential imaging modality in the characterization of metabolism within the tumor, has successfully evolved in the diagnosis, staging, and assessment of treatment response in patients with breast cancer. Cancer-associated fibroblasts (CAFs) are a crucial component of the tumor stroma with diverse functions. Fibroblast activation protein (FAP), a type II membrane-bound glycoprotein from the dipeptidyl peptidase-4 family, is highly expressed in the CAFs of several epithelial carcinomas, including breast cancer, coupled with relatively low expression in normal tissue. Gallium-68 (68Ga)-conjugated FAP inhibitor (FAPI), a new radiotracer targeting FAP, has been developed for targeting FAP and tumor-stromal visualization. With its fast renal clearance and high tumor-to-background ratio, 68Ga-FAPI has been successfully validated in multi-types of tumors. This study aims to evaluate the performance and value of 68Ga- FAPI PET/CT in patients with breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* age 18-80 years old;
* newly diagnosed BC confirmed by biopsy or with BI-RADS category 4C or 5 lesions by US or MG;
* BC clinical stagecT1-3 cN0-3 M0;
* no prior treatment for BC.

Exclusion Criteria:

* pregnancy;
* breastfeeding;
* patients who were unwilling to undergo PET/CT scans.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic Performance (1) | Through study completion, an average of 1 year
  Diagnostic performance including sensitivity, specificity, accuracy, positive predictive value and negative predictive value of 68Ga-FAPI PET/CT in the detection of ALN metastasis according to the pathological reference standard on a per-patient basis, compared with 18F-FDG PET/CT and ultrasound.

SECONDARY OUTCOMES:
Clinical Stage | Through study completion, an average of 1 year
  Clinical stage changed by 68Ga-FAPI PET/CT compared to 18F-FDG PET/CT.
Diagnostic Performance (2) | Through study completion, an average of 1 year
  Diagnostic performance of ALN metastasis of 68Ga-FAPI PET/CT with or without previous biopsy on breast lesion.
Safety | Through study completion, an average of 1 year
  Short-term adverse effects (AEs) after 68Ga-FAPI injection.

CONTACTS AND LOCATIONS:
Overall Officials: Li Huo, M.D., Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China